CLINICAL TRIAL: NCT04921969
Title: A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream Followed by a Long-Term Safety Extension Period in Children (Ages≥ 2 Years to < 12 Years) With Atopic Dermatitis ((TRuE-AD3)
Brief Title: A Study to Assess the Efficacy and Safety of Ruxolitinib Cream in Children With Atopic Dermatitis (TRuE-AD3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-305
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Ruxolitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ruxolitinib (1.5% Cream) (Experimental): Study drug will be administered twice daiily.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib (0.75% cream) (Experimental): Study drug will be administered twice daily.
  Interventions: Drug: Ruxolitinib
- Vehicle Cream (Placebo Comparator): Vehicle cream will be administered twice daily.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib — The study cream will be applied topically twice a day for up to 52 weeks.
  Other Names: Jakafi
  Arms: Ruxolitinib (0.75% cream); Ruxolitinib (1.5% Cream)
Drug: Vehicle Cream — Matching vehicle cream will be applied topically twice a day for up to 8 weeks.
  Other Names: Placebo
  Arms: Vehicle Cream

SUMMARY:
The purpose of the study is to assess the efficacy and safety of ruxolitinib cream in children with Atopic Dermatitis. This is a randomized, double-blind, Vehicle Controlled study. Participants will be randomized 2:2:1 to blinded treatment with ruxolitinib cream 0.75% ,1.5% , or vehicle cream, with stratification by baseline IGA score and age. At Week 8, efficacy will be evaluated. Participants who complete Week 8 assessments with no additional safety concerns will continue into the 44-week Long Term Safety (LTS) period with the same treatment regimen, except those initially randomized to vehicle cream will be rerandomized (1:1) in a blinded manner to 1 of the 2 active treatment groups (ruxolitinib cream 0.75% or 1.5%).

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Atopic Dermatitis (AD) as defined by the Hanifin and Rajka criteria.
* Participants with AD duration of at least 3 months (participant/parent/guardian may verbally report signs and symptoms of AD with onset at least 3 months prior).
* Participants with IGA score of 2 to 3 at the screening and baseline visits.
* Participants with %BSA (excluding scalp) of AD involvement of 3% to 20% at screening and baseline visits.
* For children aged 6 years to < 12 years, baseline itch NRS score ≥ 4.
* Participants/guardians who agree to discontinue all agents used by the participant to treat AD from the screening visit through the final safety follow-up visit.
* Participants with at least 1 target lesion that measures at least 5 cm2 at the screening and baseline visits. The target lesion must be representative of the participant's disease state but not located on the hands, feet, or genitalia.
* Willingness to avoid pregnancy or fathering a child for the duration of study participation.

Exclusion Criteria:

* An unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks before the baseline visit.
* Concurrent conditions and history of other diseases as follows:

  1. Immunocompromised
  2. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit.
  3. Active acute bacterial, fungal, or viral skin infection within 1 week before the baseline visit.
  4. Any other concomitant skin disorder, pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise participant safety.
  5. Presence of AD lesions only on the hands or feet without prior history of involvement of other classic areas of involvement such as the face or the flexural folds.
  6. Other types of eczema.
  7. Chronic asthma requiring more than 880 µg of inhaled budesonide or equivalent high dose of other inhaled corticosteroids.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Use of any of the following treatments within the indicated washout period before the baseline visit:

  1. 5 half-lives or 12 weeks, whichever is longer - biologic agents (eg, dupilumab).
  2. 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogues, cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus).
  3. 2 weeks - immunizations with activated vaccines; sedating antihistamines unless on a long-term stable regimen (nonsedating antihistamines are permitted). Note: Live vaccines are not recommended during the VC period.
  4. 1 week - use of topical treatments for AD (other than bland emollients, eg, Aveeno® creams, ointments, sprays, soap substitutes), such as corticosteroids, calcineurin inhibitors, PDE4 inhibitors, coal tar (shampoo), topical antibiotics, or antibacterial cleansing body wash/soap. Note: Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week.
* Participants who have previously received JAK inhibitors, systemic or topical. -Ultraviolet light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 2 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the participant's AD.-
* Positive serology test results at screening for HIV antibody.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the baseline visit with another investigational medication or current enrollment in another investigational drug protocol.
* In the opinion of the investigator, unable or unlikely to comply with the administration schedule and study evaluations.
* Employees of the sponsor or investigator or otherwise dependents of them.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Angel, MD, Study Director — Incyte Corporation
Locations (67):
- United States (64):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Cahaba Dermatology, Hoover, Alabama
  - Physicians Research Group Ii, Gilbert, Arizona
  - Cct Research With Center For Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - First Oc Dermatology, Fountain Valley, California
  - Iact Health, Los Angeles, California
  - Metropolis Dermatology, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Madera Family Medical Group, Madera, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Palmtree Clinical Research-Clinedge-Ppds, Palm Springs, California
  - Integrated Research of Inland, Inc, Riverside, California
  - Clinical Science Institute Clinical Research Specialists Inc, Santa Monica, California
  - Phdermatology, Clearwater, Florida
  - Life Clinical Trials Margate, Margate, Florida
  - Acevedo Clinical Research, Miami, Florida
  - Pediatric Center of Excellence Pce Miami Pediatric Endocrinology, Llc, Miami, Florida
  - The Childrens Skin Center Csc Miami, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Ciocca Dermatology Pa, Miami, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Aeroallergy Research Lab of Savannah, Savannah, Georgia
  - Northwestern Memorial Hospital-Arkes Pavilion, Chicago, Illinois
  - Sneeze Wheeze and Itch Associates Llc, Normal, Illinois
  - Northshore Medical Group Dermatology Skokie, Skokie, Illinois
  - Dermatology Specialists Research Indiana, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group Llc, Indianapolis, Indiana
  - Kansas City Dermatology P.A., Lenexa, Kansas
  - Office of Michael W. Simon, Md, Nicholasville, Kentucky
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Delricht Clinical Research-Clinedge-Ppds Baton Rouge, Baton Rouge, Louisiana
  - Delricht Research-Touro Medical Center, New Orleans, Louisiana
  - Lawrence J. Green, Md. Llc, Rockville, Maryland
  - Henry Ford Medical Center-New Center One, Detroit, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Skin Specialists Pc the Advanced Skin Research Center, Omaha, Nebraska
  - Dr Bobby Buka, Md Greenwich Village, New York, New York
  - New York University Langone Medical Center-Fink Children'S Ambulatory Care Center, New York, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Velocity Clinical Research Grants Pass Clinical Research Institute of Southern Oregon Pc, Grants Pass, Oregon
  - Cyn3Rgy Research-Clinedge-Ppds, Gresham, Oregon
  - Velocity Clinical Research-Medford, Medford, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Knight Cancer Institute At Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology Alamo Heights Office, San Antonio, Texas
  - Allergy and Asthma Care of Waco, Pa, Waco, Texas
  - Intermountain Clinical Research Icr Draper, Draper, Utah
  - Springville Dermatology, Springville, Utah
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - Skindc Clinic, Arlington, Virginia
  - Pi Coor Clinical Research Llc, Burke, Virginia
  - Clinical Research Partners Llc, Richmond, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
  - Children'S Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Dermatology Research Institute, Calgary, Alberta
  - Leader Research, Hamilton, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 330 participants were enrolled at 48 study centers in the United States and Canada.
Pre-assignment Details: Participants who completed Week 8 assessments of the Vehicle-controlled (VC) Period with no safety concerns continued in the 44-week Long-term Safety (LTS) Period. Participants who were on active treatment during the VC Period continued with the same treatment regimen in the LTS Period, and those who applied vehicle cream during the VC Period were equally randomized into 1 of the 2 active treatment groups (ruxolitinib 0.75%, ruxolitinib 1.5%) cream during the LTS Period.
Groups:
- VC Period: Vehicle Cream BID: Participants received ruxolitinib matching vehicle cream, applied topically to the affected areas as a thin film twice daily (BID) 8 hours apart from Day 1 up to Week 8. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- VC Period: Ruxolitinib 0.75% Cream BID: Participants received ruxolitinib 0.75% cream, applied topically to the affected areas as a thin film BID 8 hours apart from Day 1 up to Week 8. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- VC Period: Ruxolitinib 1.5% Cream BID: Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film BID 8 hours apart from Day 1 up to Week 8. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID: Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID: Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 0.75% Cream BID: Participants who applied ruxolitinib 0.75% cream during the VC Period, continued applying ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 1.5% Cream BID: Participants who applied ruxolitinib 1.5% cream during the VC Period, continued applying ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
Period: VC Period (Day 1 to Week 8)
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream BID | LTS Period: Ruxolitinib 1.5% Cream BID
Started | 65 | 134 | 131 | 0 | 0 | 0 | 0
Completed | 49 | 120 | 115 | 0 | 0 | 0 | 0
Not Completed | 16 | 14 | 16 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 8 | 0 | 0 | 0 | 0
Not completed — Protocol-specified Withdrawal Criterion Met | 3 | 2 | 0 | 0 | 0 | 0 | 0
Period: LTS Period (Weeks 8 to 52)
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream BID | LTS Period: Ruxolitinib 1.5% Cream BID
Started | 0 | 0 | 0 | 25 | 24 | 119 | 114
Completed | 0 | 0 | 0 | 18 | 15 | 71 | 77
Not Completed | 0 | 0 | 0 | 7 | 9 | 48 | 37
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 6 | 18 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 3 | 22 | 18
Not completed — Protocol-specified Withdrawal Criterion Met | 0 | 0 | 0 | 1 | 0 | 1 | 2
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Follow-up Not Performed per Protocol | 0 | 0 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | Total
Number analyzed (Participants) | 65 | 134 | 131 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (3.12) | 6.6 (2.83) | 6.4 (2.94) | 6.5 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 73 | 68 | 179
  Male | 27 | 61 | 63 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 37 | 75 | 68 | 180
  Black/African-American | 19 | 45 | 42 | 106
  Asian | 3 | 7 | 11 | 21
  American-Indian/Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiian/Pacific Islander | 1 | 1 | 0 | 2
  Not Reported | 0 | 1 | 1 | 2
  Black or African American and White | 2 | 2 | 2 | 6
  Mixed, Black | 1 | 0 | 0 | 1
  Captured as Hispanic or Latino in Database | 2 | 0 | 2 | 4
  Caucasian and North African | 0 | 1 | 0 | 1
  Caregiver Did Not Identify | 0 | 1 | 0 | 1
  Puerto Rican | 0 | 1 | 0 | 1
  Black and Asian | 0 | 0 | 1 | 1
  African-American/Black, Hispanic, and Caucasian/White | 0 | 0 | 1 | 1
  Portuguese | 0 | 0 | 1 | 1
  Brazilian | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 32 | 42 | 100
  Not Hispanic or Latino | 39 | 99 | 89 | 227
  Not Reported | 0 | 1 | 0 | 1
  Unknown | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: VC Period: Percentage of Participants Who Achieved Investigator's Global Assessment - Treatment Success (IGA-TS) at Week 8
Description: The IGA is an overall eczema severity rating on a 5-point scale ranging from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. The IGA-TS is defined as an IGA score of 0 (clear skin) or 1 (almost clear skin) with ≥2 grade improvement from Baseline.
Time Frame: Baseline to Week 8
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to the study. Treatment groups for this population were defined according to the treatment assignment at the time of randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 65 | 134 | 131
percentage of participants | 10.8 [4.4 to 20.9] | 36.6 [28.4 to 45.3] | 56.5 [47.6 to 65.1]
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p = 0.0001, Exact Logistic Regression — The unadjusted p-values between each treatment group and vehicle were calculated based on Exact Logistic Regression including treatment and stratification factors to test the treatment difference; Odds Ratio (OR) = 4.74, 95% CI 2-sided [1.951 to 13.315]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 10.72, 95% CI 2-sided [4.429 to 30.042]

2. Secondary Outcome: VC Period: Percentage of Participants With a ≥4-Point Improvement in Itch Numerical Rating Scale (NRS) Score From Baseline to Week 8
Description: The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity using a diary. Participants were asked to rate the itching severity because of their AD by selecting the number from 0 (no itch) to 10 (worst imaginable itch) that best described their worst level of itching in the past 24 hours.
Time Frame: Baseline to Week 8
Population: ITT Population. Only those participants who were at least 6 years of age and had a Baseline Itch NRS Score ≥4 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 37 | 80 | 76
percentage of participants | 29.7 [15.873 to 46.980] | 37.5 [26.919 to 49.035] | 43.4 [32.083 to 55.288]
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p = 0.4198, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.610 to 3.268]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.1685, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.779 to 4.174]

3. Secondary Outcome: VC Period: Percentage of Participants With a ≥4-Point Improvement in Itch NRS Score From Baseline to Day 7 (Week 1)
Description: as for outcome 2
Time Frame: Baseline to Day 7 (Week 1)
Population: ITT Population. Only those participants who were at least 6 years of age and had a Baseline Itch NRS Score ≥4 were included in the analysis. Missing Day 7 Itch scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors, Baseline, and post-Baseline Day 1 to Day 7 Itch NRS Score as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 37 | 79 | 76
percentage of participants | 11.5 | 23.5 | 28.2

4. Secondary Outcome: VC Period: Percentage of Participants With a ≥4-Point Improvement in Itch NRS Score From Baseline to Day 3
Description: as for outcome 2
Time Frame: Baseline to Day 3
Population: ITT Population. Only those participants who were at least 6 years of age and had a Baseline Itch NRS Score ≥4 were included in the analysis. Missing Day 3 Itch scores were imputed by Multiple Imputation with Fully Conditional Specification. The multiple imputation method used treatment and observed stratification factors, Baseline, and post-Baseline Day 1 to Day 7 Itch NRS Score as predicators.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 37 | 79 | 76
percentage of participants | 4.1 | 14.6 | 12.1

5. Secondary Outcome: VC Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE is defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up.
Time Frame: from Baseline up to Week 8
Population: Safety Population: all randomized participants who applied ruxolitinib cream or vehicle cream at least once. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 65 | 134 | 130
Participants | 18 | 35 | 48

6. Secondary Outcome: LTS Period: Number of Participants With Any TEAE
Description: as for outcome 5
Time Frame: From Week 8 up to Week 56
Population: LTS Evaluable Population: all participants who applied study drug at least once during the LTS Period
Measure: Count of Participants; unit: Participants
Groups:
- LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID: Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID, as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID: Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID, as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 0.75% Cream BID: Participants who applied ruxolitinib 0.75% cream during the VC Period continued applying ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID, as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 1.5% Cream BID: Participants who applied ruxolitinib 1.5% cream during the VC Period continued applying ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID, as needed from Week 8 up to Week 52. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream BID | LTS Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 25 | 24 | 119 | 114
Participants | 9 | 13 | 57 | 63

7. Secondary Outcome: VC Period: Number of Participants With Any Grade 3 or Higher TEAE
Description: A TEAE is defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up. The severity of AEs will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated; Grade 5: fatal.
Time Frame: from Baseline up to Week 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 65 | 134 | 130
Participants | 0 | 0 | 2

8. Secondary Outcome: LTS Period: Number of Participants With Any Grade 3 or Higher TEAE
Description: as for outcome 7
Time Frame: From Week 12 up to Week 56
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream BID | LTS Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 25 | 24 | 119 | 114
Participants | 0 | 0 | 3 | 3

9. Secondary Outcome: VC Period: Percentage of Participants Who Achieved IGA-TS at Weeks 2 and 4
Description: as for outcome 1
Time Frame: Baseline to Weeks 2 and 4
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 65 | 134 | 131
percentage of participants
  Week 2 | 4.6 [1.0 to 12.9] | 24.6 [17.6 to 32.8] | 35.1 [27.0 to 43.9]
  Week 4 | 12.3 [5.5 to 22.8] | 36.6 [28.4 to 45.3] | 48.1 [39.3 to 57.0]

10. Secondary Outcome: VC Period: Percentage of Participants With a ≥4-Point Improvement in Itch NRS Score From Baseline to Week 2 and 4
Description: The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity using a diary. Participants were asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best described their worst level of itching in the past 24 hours.
Time Frame: Baseline to Weeks 2 and 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 37 | 80 | 76
percentage of participants
  Week 2 | 8.1 [1.704 to 21.910] | 23.8 [14.945 to 34.578] | 23.7 [14.682 to 34.824]
  Week 4 | 10.8 [3.025 to 25.418] | 33.8 [23.553 to 45.191] | 36.8 [26.058 to 48.686]

11. Secondary Outcome: VC Period: Percentage of Participants Who Achieved Eczema Area and Severity Index 75 (EASI75) at Weeks 2, 4, and 8
Description: The EASI scoring system examines 4 areas of the body (head/neck, trunk, upper limbs, and lower limbs) and weights them for participants of ≥8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l), each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72; the severity strata are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI75 responder was defined as a participant achieving 75% or greater improvement from Baseline in EASI score.
Time Frame: Baseline to Weeks 2, 4, and 8
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 65 | 134 | 131
percentage of participants
  Week 2 | 6.2 [1.702 to 15.013] | 35.8 [27.728 to 44.556] | 43.5 [34.876 to 52.447]
  Week 4 | 12.3 [5.466 to 22.819] | 53.0 [44.178 to 61.658] | 62.6 [53.718 to 70.890]
  Week 8 | 15.4 [7.632 to 26.478] | 51.5 [42.708 to 60.210] | 67.2 [58.432 to 75.123]

12. Secondary Outcome: VC Period: Time to Achieve Itch NRS Score Improvement of at Least 2 or 4 Points
Description: The Itch NRS is a daily participant-reported measure (24-hour recall), of the worst level of itch intensity using a diary. Participants are asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours. Kaplan-Meier estimation method was used for analyses.
Time Frame: up to Week 8
Population: ITT Population. Participants who were at least 6 years of age and had a Baseline Itch NRS score ≥2 (for assessment of improvement of at least 2 points) or ≥4 (for assessment of improvement of at least 4 points), a daily Itch NRS assessment during the VC Period, and available data were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 38 | 84 | 76
days
  Improvement of at least 2 points | 6.0 [4.0 to 21.0] | 4.0 [3.0 to 5.0] | 5.0 [3.0 to 6.0]
  Improvement of at least 4 points: number analyzed (Participants) | 37 | 79 | 76
  Improvement of at least 4 points | 23.0 [13.0 to NA] — The upper limit of the 95% confidence interval was not estimable because there were too few participants with events. | 11.0 [9.0 to 20.0] | 13.0 [9.0 to 17.0]

ADVERSE EVENTS:
Time Frame: up to 60 weeks
Description: Adverse events were assessed in members of the Safety Population (all randomized participants who applied ruxolitinib cream or vehicle cream at least once) during the VC Period and in members of the LTS Evaluable Population (all participants who applied study drug at least once during the LTS Period) during the LTS Period. For participants who were on vehicle up to Week 8 and then switched to ruxolitinib, AEs are presented by the treatment they were on at onset of AE.
Groups:
- Vehicle Cream BID: Participants received ruxolitinib matching vehicle cream, applied topically to the affected areas as a thin film twice daily (BID) from Day 1 up to Week 8.
- Ruxolitinib 0.75% Cream BID: Participants received ruxolitinib 0.75% cream, applied topically to the affected areas as a thin film BID from Day 1 up to Week 8. Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52.
- Ruxolitinib 1.5% Cream BID: Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film BID from Day 1 up to Week 8. Participants who applied vehicle cream during the VC Period were randomized at Week 8 to apply ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID as needed from Week 8 up to Week 52.
Arm/Group | Vehicle Cream BID | Ruxolitinib 0.75% Cream BID | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/159 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/159 | 3/154
Other Adverse Events (participants affected / at risk) | 4/65 | 50/159 | 49/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=65) | Ruxolitinib 0.75% Cream BID (N=159) | Ruxolitinib 1.5% Cream BID (N=154)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=65) | Ruxolitinib 0.75% Cream BID (N=159) | Ruxolitinib 1.5% Cream BID (N=154)
COVID-19 (Infections and infestations) | 1 (1) | 13 (13) | 11 (11)
Nasopharyngitis (Infections and infestations) | 1 (1) | 9 (10) | 20 (23)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 9 (10) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 10 (12) | 6 (12)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 22 (30) | 23 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT04921969/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04921969/SAP_001.pdf